CLINICAL TRIAL: NCT07020741
Title: Assessing Metabolic Health With Stable Isotope Tracer Techniques in Adults With Obesity
Brief Title: Stable Isotopes- Adults With Obesity
Acronym: Si-OBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-0166; RB25064 (Other Grant/Funding Number: University of Illinois Campus Research Board)
Record Dates: First submitted 2025-05-09; First posted 2025-06-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-06

CONDITIONS: Obese Patients (BMI ≥ 30 kg/m²); Glucose Metabolism; Protein Metabolism

STUDY DESIGN:
Intervention Model Description: The study will employ a crossover model where they will complete 2 of 2 conditions, in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IAAO (Experimental): Participants will ingest a series of 6 hourly beverages containing 50% of the daily intake of 1.1g/kg/day
  Interventions: Procedure: Indispensable Amino Acid Oxidation
- SIOGTT (Experimental): Participants will consume one 75g glucose drink dissolved in 250 ml of water.
  Interventions: Procedure: Stable Isotope Oral Glucose Tolerance Test

INTERVENTIONS:
Procedure: Indispensable Amino Acid Oxidation — Participants will ingest six hourly meals designed to provide 50% of the daily intake of 1.1 g·kgLBM. Additional energy (1.5x daily resting metabolic rate), carbohydrate (55%), and fat (35%) will be provided in beverages and protein-free cookies (for palatability). The first drink will contain priming doses of NaH13CO2 (0.176 mg·kg-1), [13C]phenylalanine (1.86 mg·kg-1), [2H5]phenylalanine (0.34 mg·kg-1) with all subsequent drinks containing 1.2 mg·kg-1 [13C]phenylalanine and 0.51 mg·kg-1 [2H5]phenylalanine.
  Other Names: IAAO
  Arms: IAAO
Procedure: Stable Isotope Oral Glucose Tolerance Test — Participants will consume a 75g glucose drink dissolved in 250 ml of water enriched with [6,6_2H2]glucose and [13C6]glucose.
  Other Names: Si OGTT
  Arms: SIOGTT

SUMMARY:
In a crossover design, 8 participants will receive caloric drinks containing stable isotopes. In one arm of the study, participants will consume 6 hourly drinks containing two stable isotopes. Repeated blood, breath, urine, and muscle biopsies will be taken. In the second arm, participants will consume 1 drink containing 75g glucose, labeled with two stable isotopes of glucose. Periodic blood and breath will be taken over three hours.

DETAILED DESCRIPTION:
1. Enrollment, Informed Consent, and Screening Questionnaires (Virtual): Prior to study enrollment, participants will be asked to read a digital copy of an informed consent document provided using the e-Consent framework through the Research Electronic Data Capture (REDCap) system. Should participants have any questions about the study after reading the document, they will be encouraged to contact the research team prior to providing informed consent. Upon provision of informed consent, participants will receive an email with questionnaires designed to assess eligibility for the study through REDCap. Specifically, participants will be asked to complete a health and medical history questionnaire, physical activity readiness questionnaire (PARQ), International Physical Activity Questionnaire Long Form (IPAQ), and Godin-Shephard Leisure-Time Physical Activity Questionnaire (LTPAQ). Information from the medical history questionnaire, PARQ, and LTPAQ will be used to assess exclusion criteria and the IPAQ be used to assess baseline habitual activity level. Upon completion of these questionnaires, the research team will review responses and determine eligibility. Should Participants be eligible, researchers will work with the participant to schedule subsequent visits
2. Preliminary Testing (Visit 1): Participants will arrive for the preliminary testing session after an overnight fast.

Urine samples: 30mL of urine at time points -30 min, 0 min, 240 min, 300 min, and 360 min. Briefly, participants will be provided with a urine collection cup, alcohol wipes, and gloves and asked to fill the cup about 3/4 of they way.

Blood Collection: ~88 mL will be collected during the trial.

Breath Collection: At -30 minutes, 0 minutes, 120 minutes, 240 minutes, 300 minutes, 360 minutes, we will measure the air exhaled. To do this, participants breathe normally through a hose. Immediately after, they will exhale into a separate mouthpiece attached to a plastic bag.

Muscle Collection: A total of 2 muscle biopsies will be collected during the trial. The biopsy procedure involves removal of a small piece of muscle tissue using a sterile hollow needle (Bergström needle) and will be performed by Dr. Nicholas Burd under the auspices of Dr. Jared Willard, MD. Participants will rest on a bed and the area for the biopsy will be shaved, if required. Subsequently, the area will be sterilized using 4% chlorhexidine gluconate before 5 mL of local anesthetic (2% Xylocaine with 1:100,000 epinephrine) is injected subcutaneously with special care to avoid infiltrating the muscle. Once the anesthetic is active, a small incision will be made in the skin in order to create an opening through which to put the biopsy needle for tissue collection. Dr. Burd will quickly cut of a small piece of muscle. the subjects may feel a sensation of deep pressure in their leg. A sterile disposable drape will be placed under the participant's thigh and sterile gloves will be used for all biopsy procedures.

After the biopsy is completed, a trained research team member will apply pressure with sterile gauze until the bleeding stops (at least 15 minutes). Subsequently, the incision site will be closed using butterfly stitches (Steri-strips) following by application of a bandage. An elastic pressure wrap will be applied on top of the bandage in order to minimize the chance of bruising. Participants will then be instructed to leave the butterfly stitches and the pressure wrap on the wound for 96 and 24 hrs, respectively.

The participant will be provided with a "biopsy care kit" (described in section 10.1/Biopsy care kit) in order to properly care for the incision after leaving the laboratory. A member of the research team will contact the participants in the day following the trial to check on the healing process.

After blood, breath, and muscle samples of time 0, participants will drink the first of a series of drinks containing [13C]phenylalanine and [2H5]phenylalanine at a ratio of 1:10 with a 1:10 ratio of total tracer to tracee (naturally occurring phenylalanine) The first drink will be primed with NaH13CO2 (0.176 mg/kg) in addition to [13C]phenylalanine and [2H5]phenylalanine mixture. Drinks will be consumed every 30 minutes for the duration of the procedure.

These drink will also contain 1.2x estimated RMR calories (divided into 12 drinks)

VCo2: Carbon dioxide production (VCO2) will be determined from expired air sampled by open circuit spirometry using an on-line, computer-based acquisition system. Participants will breathe through a one-way, high velocity non-rebreathing valve. The volume of expired air is measured by a gas flow meter. The carbon dioxide concentrations of expired air are assessed by a carbon dioxide analyser. Analog data from the gas analyser and flow meter is digitized and sent to an IBM compatible PC for calculation of VCO2 converted to Standard Temperature and Pressure Dry. Immediately after VCO2 analysis is performed (5 min), subjects are asked to exhale into a separate mouthpiece attached to a plastic bag. This particular breath sample is stored in a sterile vacutainer for future analysis of stable isotope tracer enrichment in the breath. The measurement of carbon dioxide production (VCO2) and the measurement of tracer enrichment in the breath allow us to assess how much of the protein is used for energy, rather than for building skeletal muscle proteins. Subjects are not expected to experience any discomfort from this procedure, nor will it influence their physical well-being.

(Visit 4) Stable Isotope OGTT: within 7 days after the first trail participants will be asked to return to the lab for a second procedure.

Blood Collection: Blood collection procedures will be exactly as described above. There will be a total of 9 blood collections (time -10, 10, 20, 30, 60. 90, 120, 150, 180) minutes Breath Collection: Breath collection procedures will be exactly as described above. There will be a total of 9 breath collections (-10, 10, 20, 30, 60, 90, 120, 150, 180) minutes After the blood and breath collection for time -10 minutes, participants will be asked to consume a 75 g Glucose Drink dissolved in 250 ml of water enriched with [6,6_2H2]glucose and [13C6]glucose. As stated above, blood and breath samples will be taken periodically over the next 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* ages 19-59
* Obese >/= 30 kg/m^2 and >/= 102 cm for males and >/= 88 cm for females
* Godin Leisure-time or exercise questionnaire <14 units

Exclusion Criteria:

1. Pregnant or become pregnant
2. Any known food allergies
3. Smoker
4. Are physically active
5. Have any known metabolic diseases
6. Have been weight unstable within the last 6 months (lost or gained >10% of body mass)
7. Non eumenorrheic or on a hormonal birth control

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Define obesity-related whole body protein efficiency based of the IAAO method | 0 - 6 hours observational period ingesting six hourly meals, within 1 week of preliminary testing. Baseline measures taken at --30 minutes.
  Amino Acid Oxidation of phenylalanine will be measured using the IAAO method by periodic ingestion of amino acid mixture. Trials will start at ~7:00 am (-30 minutes) with a total duration of 6.5 hours (390 minutes) Measurements of breath (-30, 0, 120, 240, 270, 300, 330 and 360 minutes), Urine (-30, 0, 240, 300, and 360 minutes), muscle biopsy (-30 and 360 minutes) and blood (-30, 0, 30, 60, 90,120, 180, 240, 300, and 360 minutes) will be used to determine the whole body efficiency of protein in obese populations.
Assessment of oral glucose tolerance based on a dual tracer technique | 0- 3 hour observational period. Within 1 week of the prospective arm. Baseline taken at -30 minutes.
  Measure glucose kinetics via [13C] and D5 Glucose over 3 hours to determine glucose tolerance. Trials will start at ~7:00 am (-10 minutes) and last ~ 3 hours. (190 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Freer Hall - University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Because it is not planned to published in any ICMJE journal.